CLINICAL TRIAL: NCT00070070
Title: NY-ESO-1 Protein Immunization of Post-Cystectomy or Post-Nephroureterectomy Patients With Transitional Cell Carcinomas
Brief Title: Vaccine Therapy in Treating Patients With Transitional Cell Carcinomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LUD2002-004; MSKCC-03047 (Other: MSKCC); LUDWIG-LUD2002-004 (Other: Ludwig Institute for Cancer Research); CDR0000329920 (Other: Ludwig Institute for Cancer Research)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Transitional Cell Carcinoma
Keywords: Bladder cancer; Renal pelvis cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — BCG Vaccine; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: This study was open-label, and eligible patients were sequentially entered at the time they presented in clinic. Patients were sequentially assigned to one of four groups according to HLA-A2 characteristic and previous Bacille Calmette Guerin (BCG) therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): HLA-A2 Status Positive, Previous BCG Therapy; All patients underwent skin testing with the purified protein derivative (PPD) test.
  NY-ESO-1 protein, 75 mcg, was administered by intradermal injection every week for 6 weeks. TICE®-strain BCG, 1 x 10E6 viable units in Purified Protein Derivative (PPD) negative patients and 1 x 10E5 viable units in PPD positive (induration greater than or equal to 10 mm) patients, were mixed with each protein vaccination for the first 2 weeks only. For the last 4 weeks GM-CSF, 100 mcg, was mixed with NY-ESO-1 protein given once a week for 4 weeks, intradermally. GM-CSF alone was given subcutaneously on the day prior to the administration of the co-mixture (NY-ESO-1 Protein/GM-CSF) and for 3 days after.
  Interventions: Biological: TICE®-strain BCG; Biological: NY-ESO-1 protein; Biological: sargramostim
- Cohort 2 (Experimental): HLA-A2 Status Positive, No Previous BCG Therapy; All patients underwent skin testing with the purified protein derivative (PPD) test.
  NY-ESO-1 protein, 75 mcg, was administered by intradermal injection every week for 6 weeks. TICE®-strain BCG, 1 x 10E6 viable units in Purified Protein Derivative (PPD) negative patients and 1 x 10E5 viable units in PPD positive (induration greater than or equal to 10 mm) patients, were mixed with each protein vaccination for the first 2 weeks only. For the last 4 weeks GM-CSF, 100 mcg, was mixed with NY-ESO-1 protein given once a week for 4 weeks, intradermally. GM-CSF alone was given subcutaneously on the day prior to the administration of the co-mixture (NY-ESO-1 Protein/GM-CSF) and for 3 days after.
  Interventions: Biological: TICE®-strain BCG; Biological: NY-ESO-1 protein; Biological: sargramostim
- Cohort 3 (Experimental): HLA-A2 Status Negative, Previous BCG Therapy; All patients underwent skin testing with the purified protein derivative (PPD) test.
  NY-ESO-1 protein, 75 mcg, was administered by intradermal injection every week for 6 weeks. TICE®-strain BCG, 1 x 10E6 viable units in Purified Protein Derivative (PPD) negative patients and 1 x 10E5 viable units in PPD positive (induration greater than or equal to 10 mm) patients, were mixed with each protein vaccination for the first 2 weeks only. For the last 4 weeks GM-CSF, 100 mcg, was mixed with NY-ESO-1 protein given once a week for 4 weeks, intradermally. GM-CSF alone was given subcutaneously on the day prior to the administration of the co-mixture (NY-ESO-1 Protein/GM-CSF) and for 3 days after.
  Interventions: Biological: TICE®-strain BCG; Biological: NY-ESO-1 protein; Biological: sargramostim
- Cohort 4 (Experimental): HLA-A2 Status Negative, No Previous BCG Therapy; All patients underwent skin testing with the purified protein derivative (PPD) test.
  NY-ESO-1 protein, 75 mcg, was administered by intradermal injection every week for 6 weeks. TICE®-strain BCG, 1 x 106 viable units in Purified Protein Derivative (PPD) negative patients and 1 x 105 viable units in PPD positive (induration greater than or equal to 10 mm) patients, were mixed with each protein vaccination for the first 2 weeks only. For the last 4 weeks GM-CSF, 100 mcg, was mixed with NY-ESO-1 protein given once a week for 4 weeks, intradermally. GM-CSF alone was given subcutaneously on the day prior to the administration of the co-mixture (NY-ESO-1 Protein/GM-CSF) and for 3 days after.
  Interventions: Biological: TICE®-strain BCG; Biological: NY-ESO-1 protein; Biological: sargramostim

INTERVENTIONS:
Biological: TICE®-strain BCG
  Other Names: BCG Live; Tice® BCG; BCG Vaccine
Biological: NY-ESO-1 protein
Biological: sargramostim
  Other Names: GM-CSF

SUMMARY:
RATIONALE: Vaccines made from peptides may make the body build an immune response to kill tumor cells. Biological therapies, such as Bacille Calmette Guerin (BCG) and sargramostim (GM-CSF), use different ways to stimulate the immune system and stop tumor cells from growing. Combining vaccine therapy with biological therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects of giving vaccine therapy together with BCG and sargramostim in treating patients who have undergone cystectomy for transitional cell carcinomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of NY-ESO-1 peptide vaccine, Bacille Calmette Guerin (BCG), and sargramostim (GM-CSF) in post-cystectomy patients with transitional cell carcinoma of the bladder expressing NY-ESO-1 or LAGE-1 antigen.
* Determine the immunological profile (NY-ESO-1 antibody, CD8+ cells, and delayed-type hypersensitivity) induced by this regimen in these patients.

OUTLINE: This is an open-label, pilot study.

Patients receive NY-ESO-1 protein vaccine mixed with BCG intradermally (ID) once weekly on weeks 1 and 2. Patients then receive NY-ESO-1 protein mixed with sargramostim (GM-CSF) ID once weekly on day 2 of weeks 3-6. Patients also receive GM-CSF subcutaneously alone on days 1, 3, 4, and 5 of weeks 3-6.

ELIGIBILITY:
Inclusion Criteria

1. Post-cystectomy or post-nephroureterectomy patients with histological confirmation of transitional cell carcinoma.
2. Patients must have had a cystectomy or nephroureterectomy within 16 weeks of first vaccination.
3. At least 4 weeks since surgery prior to receiving the first vaccination.
4. Radiological imaging to document no evidence of disease within one month prior to receiving the first vaccination.
5. Laboratory values within the following limits:

Hemoglobin ≥ 10.0 g/dL Neutrophil count ≥ 1.5 x 10E9/L Lymphocyte count ≥ 0.5 x 10E9/L Platelet count ≥ 100 x 10E9/L Serum creatinine ≤ 1.8 mg/dL Serum bilirubin ≤ 2mg/dL Serum aspartate aminotransferase (AST) (SGOT) <2.5 X ULN Serum alanine aminotransaminase (ALT) (SGPT) <2.5 X ULN 6. Performance status ≤ 2 (ECOG Scale) and life expectancy ≥ 3 months. 7. Age ≥ 18 years. 8. Fertile patients must have a negative urine or serum pregnancy test and use barrier method contraception before, during and for 6 months after protocol therapy. Patients are encouraged to continue barrier method contraception for two years or longer after treatment.

9. Able and willing to give valid written informed consent. Exclusion Criteria

1. Clinically significant heart disease (NYHA Class III or IV).
2. Presence of severe reaction to PPD (purified protein derivative) (>40 mm induration).
3. Prior malignancy within 5 years that has been treated with extensive chemotherapy / radiation therapy and have the potential for immune dysfunction or who have evidence of metastasis at the time of registration.
4. Other serious illnesses, e.g., serious infections requiring antibiotics, bleeding disorders, antibiotic use within 5 days of treatment.
5. Previous bone marrow or stem cell transplant.
6. History of immunodeficiency disease or autoimmune disease.
7. Known positive HIV test.
8. Chemotherapy, radiation therapy, or immunotherapy within 4 weeks before study entry (6 weeks for nitrosoureas).
9. Concomitant treatment with corticosteroids (within 30 days of enrollment and during treatment), antihistaminic drugs, or nonsteroidal anti-inflammatory drugs (unless chronically used in low doses for prevention of an acute cardiovascular event or pain control). Topical or inhalational steroids are permitted.
10. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to enrollment.
11. Mental disorders that may compromise the ability to give informed consent and comply with the requirements of the study.
12. Lack of availability of the patient for immunological and clinical follow-up assessment.
13. Positive urine or serum pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2003-10-28 (Actual); Primary Completion 2006-01-03 (Actual); Study Completion 2013-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean F. Bajorin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Harry W. Herr, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sharma P, Bajorin DF, Jungbluth AA, Herr H, Old LJ, Gnjatic S. Immune responses detected in urothelial carcinoma patients after vaccination with NY-ESO-1 protein plus BCG and GM-CSF. J Immunother. 2008 Nov-Dec;31(9):849-57. doi: 10.1097/CJI.0b013e3181891574. PMID 18833002

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 4: HLA-A2 Status Negative, No Previous BCG Therapy; All patients underwent skin testing with the purified protein derivative (PPD) test.
  NY-ESO-1 protein, 75 mcg, was administered by intradermal injection every week for 6 weeks. TICE®-strain BCG, 1 x 10E6 viable units in Purified Protein Derivative (PPD) negative patients and 1 x 10E5 viable units in PPD positive (induration greater than or equal to 10 mm) patients, were mixed with each protein vaccination for the first 2 weeks only. For the last 4 weeks GM-CSF, 100 mcg, was mixed with NY-ESO-1 protein given once a week for 4 weeks, intradermally. GM-CSF alone was given subcutaneously on the day prior to the administration of the co-mixture (NY-ESO-1 Protein/GM-CSF) and for 3 days after.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 1 | 0 | 0 | 5
Completed | 1 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 1 | 0 | 0 | 5 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 0 | 1
  >=65 years | 0 | 0 | 0 | 5 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 1
  Male | 1 | 0 | 0 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 0 | 5 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 0 | 0 | 5 | 6
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  |  | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: All adverse events were graded according to the National Cancer Institute Common Toxicity Criteria (CTCAE) (Version 3.0). A Dose limiting toxicity (DLT) was defined as:
  * ≥ Grade 2 autoimmune phenomena
  * Asymptomatic bronchospasm or generalized urticaria
  * ≥ Grade 3 hematological and non hematological toxicities. To be dose limiting, an adverse event must have been definitely, probably, or possibly related to the administration of the study treatment. Patients who experienced a DLT were removed from study.
Time Frame: up to 12 weeks
Population: All participants who received at least one study treatment. One participant in Cohort 4 did not have HLA-A2 status tested.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 1 | 0 | 0 | 5
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Patients Developing NY-ESO-1 Antibodies After Treatment
Description: Blood samples were obtained at baseline, and at weeks 2, 4, 6, 8 and 12 for the assessment of NY-ESO-1 and LAGE-1 specific antibodies by enzyme-linked immunosorbent assay (ELISA).
Time Frame: up to 12 weeks
Population: All participants who received study therapy and had blood samples taken for antibody analysis before and after treatment. One participant in Cohort 4 did not have HLA-A2 status tested.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 1 | 0 | 0 | 5
Participants
  Number of Participants with NY-ESO-1 Antibodies at Baseline and After Treatment | 1 | 0 | 0 | 0
  Number of Participants with No NY-ESO-1 Antibodies at Baseline and Antibodies After Treatment | 0 | 0 | 0 | 4
  Number of Participants with No NY-ESO-1 Antibodies at Baseline and No Antibodies After Treatment | 0 | 0 | 0 | 1

3. Secondary Outcome: Number of Patients With CD4+ and CD8+ T-cell Responses.
Description: Blood samples were obtained at baseline, and at weeks 2, 4, 6, 8 and 12 for the assessment of NY-ESO-1 specific T-cell responses by ELISPOT. T-cell responses were monitored after in vitro sensitization with either overlapping peptides from NY-ESO-1 or recombinant adenovirus encoding NY-ESO-1 (adeno-NY-ESO-1), and with control peptides or recombinant vectors encoding Influenza-derived proteins.
Time Frame: up to 12 weeks
Population: All participants who received at least one dose of study therapy and had pre- and post-treatment samples taken for analysis. One participant in Cohort 4 did not have HLA-A2 status tested.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 1 | 0 | 0 | 5
Participants
  CD4+ T-Cell Responses: Number of Participants with Responses | 1 | 0 | 0 | 5
  CD4+ T-Cell Responses: Number of Participants without Responses | 0 | 0 | 0 | 0
  CD8+ T-Cell Responses: Number of Participants with Responses | 0 | 0 | 0 | 1
  CD8+ T-Cell Responses: Number of Participants without Responses | 1 | 0 | 0 | 4

4. Secondary Outcome: Delayed-type Hypersensitivity (DTH) as Measured by the Number of Participants With Induration and/or Redness at Each Timepoint
Description: NY-ESO-1-specific DTH skin reaction was measured at baseline and weeks 3 and 8.The peptide solution (10 μg peptide in 0.1ml normal saline) was injected intradermally at a separate site from the vaccination to give a visible and palpable skin depot. Assessment of DTH reactions was performed 48 h after injection.
  The extent and intensity of DTH reactions was documented by measuring visible "redness", palpable "induration" and other signs of local skin irritation or necrosis.
Time Frame: up to 8 weeks
Population: All participants who received at least one dose of study treatment and received the DTH test at the respective timepoint. One participant in Cohort 4 did not have HLA-A2 status tested.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 1 | 0 | 0 | 5
Participants
  Baseline: Number of Participants with Induration and/or Redness | 0 | 0 | 0 | 2
  Baseline: Number of Participants with No Induration and/or Redness | 1 | 0 | 0 | 3
  Week 3: number analyzed (Participants) | 1 | 0 | 0 | 4
  Week 3: Number of Participants with Induration and/or Redness | 0 | 0 | 0 | 2
  Week 3: Number of Participants with No Induration and/or Redness | 1 | 0 | 0 | 2
  Week 8: number analyzed (Participants) | 1 | 0 | 0 | 4
  Week 8: Number of Participants with Induration and/or Redness | 0 | 0 | 0 | 1
  Week 8: Number of Participants with No Induration and/or Redness | 1 | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Description: All AEs occurring during the study were to be documented in the source records and on the respective Case Report Form Adverse Event page, regardless of the assumption of a causal relationship. All events, which occurred after signed informed consent, were to be documented. Toxicity was evaluated according to the National Cancer Institute CTCAE Version 3.0.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/0 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0 | 0/5
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/0 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=1) | Cohort 2 (N=0) | Cohort 3 (N=0) | Cohort 4 (N=5)
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 0 | 5
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Peripheral edema (Cardiac disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No